CLINICAL TRIAL: NCT03380702
Title: Influence of Tooth Whitening on Changes in Quality of Life: a Randomized Double-blinded Placebo-controlled Trial
Brief Title: Influence of Tooth Whitening on Changes in Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Kovacevic Pavicic (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Sponsor-Investigator, Daniela Kovacevic Pavicic, professor, University of Rijeka
Organization: University of Rijeka (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2170-24-01-15-04
Record Dates: First submitted 2017-11-22; First posted 2017-12-21 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Tooth Discoloration; Quality of Life
Keywords: colour; dental aesthetics; perceptions; quality of life; tooth whitening
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: RANDOMIZED DOUBLE-BLINDED PLACEBO-CONTROLLED TRIAL
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whitening photoactivation gel (Active Comparator): exposure to hydrogen gel and photoactivation for teeth whitening
  Interventions: Procedure: whitening photoactivation gel
- placebo (Placebo Comparator): exposure to gel without active whitening substance and the same photoactivation source as active comparator
  Interventions: Procedure: placebo

INTERVENTIONS:
Procedure: whitening photoactivation gel — 35 subjects in active comparator group
  Arms: whitening photoactivation gel
Procedure: placebo — 35 subjects in placebo comparator group
  Arms: placebo

SUMMARY:
Lighter tooth color may improve patient satisfaction with facial aesthetics. Few data exist regarding the impact and association of of tooth color connection with quality of life.The purpose of this research is to explore the extent to which patients perceive a color change and difference in quality of life induced by tooth whitening after one week and after one year.

A plan is to assess 100 participants for eligibility (aged 18-30 years) and to enroll at least 70 and randomly assign to an active or a control group (equal number of participans in each group). Their anterior teeth in both jaws will be bleached with a photo-activated whitening gel, or will be subjected to a placebo. Lightness, chroma and translucency of teeth will be assessed before (T0), one week (T1) and one year (T2) after the procedure by a spectrophotometer. The subjects in both occasions will administrate the psychometric instrumetns Psychosocial Impact of Dental Aesthetics Questionnaire, Orofacial Esthetic Scale, Oral Health Impact Profile and Smile Esthetics Related Quality of Life. Influence of personality traits on the perception of changes in smile aesthetics and qualiy of life will be also explored (extraversion, conscientiousness, neuroticism, agreeableness, openness to experience, perfectionism, self-esteem, body image).

DETAILED DESCRIPTION:
The aim of the trial is to explore influence of teeth whitening on the perception of dentofacial aesthetics. Influence of personality traits on this relationship is also to be explored (extraversion, conscientiousness, neuroticism, agreeableness, openness to experience, perfectionism, self-esteem, body image). All total of 70 examinees (young adults) at baseline (T0) will administrate psychometric instruments Oral Health Impact Profile (OHIP), Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ), Orofacial Esthetic Scale (OES), Smile esthetics related quality of life (SERQoL), Big Five Inventory (BFI), Rosenberg's Self-Esteem Scale (RSS), Frost Multidimensional Perfectionism Sale (FMPS), and a newly developed short form instruments for body image, perfectionism, self-esteem and perception of body appearance. The elements of tooth color (lightness, chroma and translucency) will be assessed by spectrophotometer (SpectroShade, MHT, Italy) at baseline (T0), after one week (T1) and after one year (T2). The precision and accuracy of the instrument will be checked by repeated measurements and by comparison with the gold standard. Examinees will be randomly assigned to the active or control group using the "random between" function in Microsoft Excell. Teeth of half of subjects will be bleached using a lamp and photo-activated bleaching gel (Signal Easy Lamp Plus and Signal Fast Professional plus set, Signal, Unilever, Argentina), while the remaining half will be subjected to a placebo, i.e. a gel without active substance.

After one week (T1) the elements of tooth color will be assessed again and color change will be calculated (ΔE). Pain induced by whitening procedure will be assessed by using 10mm visual analogue scale. Participants will administrate instruments OHIP, PIDAQ, OES, SERQoL and short form instruments for body image, perfectionism, self-esteem and perception of body appearance. A year after the whitening procedure (T2) the elements of toth color will be assessed again and the same instruments as in T1 will be administrated. The short-term (T0-T1) and long-term (T0-T2) effect of teeth whitening on the changes in perception of dentofacial aesthetics and quality of life is to be analyzed.

The results will be analysed by using t-test, analysis of variance and covariance, and Pearson correlations.

ELIGIBILITY:
Inclusion Criteria:

* presence of a complete anterior tooth segment free of caries
* anterior tooth segment free of fillings
* anterior tooth segment free of prosthetic restorations

Exclusion Criteria:

* Gingivitis present
* Malocclusion present (Index of Orthodontic Treatment Need-Dental Health Component ≤3 and Aesthetic Component ≤4)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
change from baseline color at one week | one week after whitening
  change of color of teeth (ΔE) by spectrophotometer in scalar points (range 1-10)
change from baseline color at one year | one year after whitening
  change of color of teeth (ΔE) by spectrophotometer in scalar points (range 1-10)
change from psychosocial impact of dental aesthetics at one week | one week after whitening
  psychosocial impact of dental aesthetics measured by Psychosocial impacr of dental aesthetics questionnaire (PIDAQ; scalar points, range 0-32)
change from psychosocial impact of dental aesthetics at one year | one year after whitening
  psychosocial impact of dental aesthetics measured by Psychosocial impacr of dental aesthetics questionnaire (PIDAQ; scalar points, range 0-32)
change from baseline smile esthetics related quality of life at one week | one week after whitening
  smile esthetics related quality of life measured by Smile esthetics related quality of life quaetionnaire (SERQoL; scalar points, range 4-20)
change from baseline smile esthetics related quality of life at one year | one year after whitening
  smile esthetics related quality of life measured by Smile esthetics related quality of life quaetionnaire (SERQoL; scalar points, range 4-20)
change from baseline satisfaction with orofacial aesthetics at one week | one week after whitening
  satisfaction with orofacial aesthetics measured by Orofacial esthetic scale (OES; scalar points, range 1-45)
change from baseline satisfaction with orofacial aesthetics at one year | one year after whitening
  satisfaction with orofacial aesthetics measured by Orofacial esthetic scale (OES; scalar points, range 1-45)
change from baseline oral health-related quality of life at one week | one week after whitening
  oral health-related quality of life measured by Oral health impact profile instrument (OHIP; scalar points, range 0-56)
change from baseline oral health-related quality of life at one year | one year after whitening
  oral health-related quality of life measured by Oral health impact profile instrument (OHIP; scalar points, range 0-56)

SECONDARY OUTCOMES:
change from baseline lightness at one week | one week after whitening
  lightness of teeth measured by spectrophotometer (scalar range 67-83)
change from baseline lightness at one year | one year after whitening
  lightness of teeth measured by spectrophotometer (scalar range 67-83)
change from baseline chroma at one week | one week after whitening
  chroma of teeth measured by spectrophotometer (range 11-25)
change from baseline chroma at one year | one year after whitening
  chroma of teeth measured by spectrophotometer (range 11-25)
change from baseline translucency at one week | one week after whitening
  transluceny of teeth measured by spectrophotometer (range 0-13)
change from baseline translucency at one year | one year after whitening
  transluceny of teeth measured by spectrophotometer (range 0-13)
discomfort with teeth whitening | one week after whitening
  discomfort with teeth whitening assessed by visual-analogue scale (scalar ponts 1-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical faculty University of Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No
The publication of scientific manuscript.

REFERENCES:
- [Background] Kovacevic Pavicic D, Pavlic A, Kinkela Devcic M, Lajnert V, Spalj S. Tooth Color as a Predictor of Oral Health-Related Quality of Life in Young Adults. J Prosthodont. 2019 Apr;28(4):e886-e892. doi: 10.1111/jopr.12666. Epub 2017 Oct 31. PMID 29086473
- [Derived] Batinic M, Kovacevic Pavicic D, Sango A, Brumini M, Spalj S. Effect of personality characteristics on perception of tooth whitening outcome in young adults in long-term: a randomised, double-blind, placebo controlled trial. Head Face Med. 2025 Aug 7;21(1):57. doi: 10.1186/s13005-025-00536-3. PMID 40775639
- [Derived] Kovacevic Pavicic D, Kolceg M, Lajnert V, Pavlic A, Spalj S. Changes in quality of life induced by tooth whitening are not influenced by global self-esteem: a randomized double-blind placebo-controlled trial. Odontology. 2020 Jan;108(1):143-151. doi: 10.1007/s10266-019-00442-6. Epub 2019 Jul 9. PMID 31289971